CLINICAL TRIAL: NCT07323394
Title: Real-World Study on the Impact of Atopic Dermatitis From a Caregiver Perspective
Status: Not yet recruiting | Type: Observational
Sponsor: PeriPharm (Other)
Responsible Party: Sponsor
Other Study IDs: PROxy96AD
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis; Eczema Atopic Dermatitis; Eczema; Caregiver; Burden
Keywords: atopic dermatitis; quality of life; real-world
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregiver of child with atopic dermatitis: Caregiver of a child aged ≥2 to ≤11 years with mild to moderate atopic dermatitis
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No specific intervention is assess in this study. Observational cohort.

SUMMARY:
This study will address this gap by providing comprehensive data on disease burden from a caregiver perspective in a Canadian population, ultimately supporting improved clinical decision-making and healthcare resource allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Caregiver of a child aged ≥2 to ≤11 years with mild to moderate atopic dermatitis;
3. Able to read and understand French or English;
4. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Caregivers whose child has been diagnosed with severe atopic dermatitis ;
2. Caregivers whose child is currently treated with oral or topical Janus Kinase Inhibitor);
3. Caregivers whose child is currently participating in a clinical trial for atopic dermatitis;
4. Other parent or caregiver within the household of the child with atopic dermatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregiver of a child aged ≥2 to ≤11 years with mild to moderate atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To estimate work productivity loss in caregivers of children with mild or moderate atopic dermatitis. | At recruitment
  Using the Work Productivity and Activity Impairment questionnaire. This questionnaire provides a quantitative measure of impairment over the last 7 days and includes four metrics: absenteeism (work time missed because of health issues during the past 7 days), presenteeism (impairment while working due to health issues during the past 7 days), overall work productivity loss (combination of absenteeism and presenteeism), and activity impairment.

SECONDARY OUTCOMES:
To estimate family burden of mild to moderate atopic dermatitis in children, as reported by caregivers | At recruitment
  The Dermatitis Family Impact (DFI) questionnaire will be administered to caregivers to evaluate the family burden of pediatric atopic dermatitis. The DFI is a validated, 10-item instrument specifically developed for atopic dermatitis, covering domains such as housework, feeding, sleep, leisure activities, time spent shopping, expenditure, physical fatigue, emotional distress, relationships, helping with treatment, with a 7-day recall period. Each item is scored on a 4-point Likert scale ("Not at all = 0" to "Very much = 3"), with higher total scores indicating greater impact

IPD SHARING:
Plan to Share IPD: No